CLINICAL TRIAL: NCT01216254
Title: Prospective, Randomized Clinical Trial Comparing Pain Sensation, Seroma Formation and Quality od Life Following BCT With SLND in Breast Cancer Patients Operated With Classic Versus High-frequency Electrocoagulation.
Brief Title: Clinical Trial Comparing Outcomes of Breast Conserving Operations With Classic v High-frequency Electrocoagulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Jacek Zielinski, Assistant Profesor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKEBN/219/2010
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage 2; breast conserving therapy; sentinel lymph node dissection; high frequency electrocoagulation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Classic electrocoagulation (Active Comparator): Arm of the study where the classic low-frequency electrocoagulation is used during the operation
  Interventions: Device: classic v high-frequency electrocoagulation
- High Frequency electrocoagulation (Experimental): Arm of the study where the tested high-frequency electrocoagulation is used during the operation
  Interventions: Device: classic v high-frequency electrocoagulation

INTERVENTIONS:
Device: classic v high-frequency electrocoagulation — During the BCT with SLND the investigators would use two types of electrocoagulation. The steps of the operation would remain the same in both arms, nevertheless the tool used would vary.
  Other Names: Ellmann

SUMMARY:
The aim of this study is to assess the outcomes of breast conserving therapy operation depending on the type of surgical tool used: classic electrocoagulation with higher operative temperatures and high frequency electrocoagulation with lower operative temperatures. The investigators would assess the pain levels, length and amount of the lymphatic secretion as well as quality of life following breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18-100
* breast cancer
* stage IIA and II B (cT1a-3; cN0-1; cM0)
* no previous breast surgery
* no previous cancer
* obtained informed consent

Exclusion Criteria:

* stages I, III, IV
* localised breast infection
* previous breast surgery for any cause
* previous cancer
* no voluntary consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Pain Control | From the day before surgery up to 12 weeks (+/-2days) after surgery
  Pain assessment would be performed using Visual Analogue Scale (VAS) at the days 1-5, 10 (+/- 2), 20 (+/- 2), 30 (+/- 2), and 12 weeks (+/- 2 days). SF - MPQ questionnaire would be filled in on admission, 10th (+/- 2) post-operative day and 12 weeks (+/- 2 days)after surgery.

SECONDARY OUTCOMES:
Quality of life (QoL) | From the day before surgery up to 12 weeks (+/-2days) after surgery
  Pre-operative assessment of QoL would be performed by psychologist using questionnaires: CISS, HADS - M, Eysencka. Postoperative assessment of QoL would be performed using QLQ C30 and QLQ BR 23 questionnaires 12 weeks (+/- 2 days)after surgery
Length of lymphatic secretion | From the day before surgery up to 12 weeks (+/-2days) after surgery
  Number of days of lymphatic secretion would be assessed.
Amount of lymphatic secretion | From the day before surgery up to 12 weeks (+/-2days) after surgery
  Amount of lymphatic secretion would be measured until it stops on daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Zielinski, M.D., Ph.D., Principal Investigator — Medical University of Gdansk; Janusz Jaskiewicz, M.D., Ph.D., Study Director — Medical University of Gdansk
Locations (1):
- Department of Surgical Oncology, Gdansk, Pomeranian Voivodeship, Poland